CLINICAL TRIAL: NCT00780533
Title: Changes in and Determinants of Movement Performance, Functional Status, and Health-Related Quality of Life After Stroke Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Keh-chung Lin, Organization: School of Occupational Therapy, College of Medicine, National Taiwan University
Other Study IDs: 200712088R
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Stroke; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
A total of 144 stroke patients 6 -24 months post onset who are between 45 and 75 years old will be recruited. A randomized-blocks pretest and posttest control group design will be applied. Four groups will be involved in this project and the subjects will be stratified on two variables: impairment level of the hand and side of lesion. Randomization will be done in blocks of six and each block randomization scheme is within each stratum. Treatment regimens will be designed to ensure that patients in 4 groups receive equivalent intensity of treatment (5 days/week for 1.5 hours/day for 4 consecutive weeks) directly supervised by senior occupational therapists.

Brain and movement reorganization will be evaluated with fMRI and kinematic instrument, respectively before and after the 4-week intervention period. Clinical measures on motor impairment, daily function and quality of life will be assessed before, immediately and six months after intervention. Two examiners blind to group allocation will collaborate to provide both fMRI and kinematic evaluations and one of them will administer clinical measures. Before being allowed to work with subjects, the examiner competence will be assessed by principle investigator and co-principle investigators. Multivariate analyses of covariance will be used to examine change in brain activation, kinematic variables and clinical measures as a function of intervention while controlling for pretest data, age and onset post stroke. Multiple regression models will be established to examine the possible predictor(s) for functional outcome of each rehabilitation approach. Canonical correlation analyses will be conducted to quantify the relationship between brain/motor reorganization and clinical measures.

ELIGIBILITY:
Inclusion Criteria:

1. able to reach Brunnstrom stage III or above for the proximal part of the affected upper limb(Brunnstrom, 1970);
2. considerable nonuse of the affected upper limb (amount-of-use [AOU] score < 2.5 on the MAL) (Taub, Miller, Novack, et al. ,1993);
3. no serious cognitive deficits (score > 24 on the Mini Mental-State Exam) (Folstein, Folstein, & McHugh, 1975);
4. no balance problems compromising safety when wearing the constraint device; and,
5. no excessive spasticity (Modified Ashworth Scale ≤ 2 at any joint of the upper limb) (Bohannon, & Smith, 1987).

Ages: 50 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a group of stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chuang LL, Lin KC, Wu CY, Chang CW, Chen HC, Yin HP, Wang L. Relative and absolute reliabilities of the myotonometric measurements of hemiparetic arms in patients with stroke. Arch Phys Med Rehabil. 2013 Mar;94(3):459-66. doi: 10.1016/j.apmr.2012.08.212. Epub 2012 Sep 4. PMID 22960277
- [Derived] Chuang LL, Wu CY, Lin KC. Reliability, validity, and responsiveness of myotonometric measurement of muscle tone, elasticity, and stiffness in patients with stroke. Arch Phys Med Rehabil. 2012 Mar;93(3):532-40. doi: 10.1016/j.apmr.2011.09.014. Epub 2012 Jan 4. PMID 22222143